CLINICAL TRIAL: NCT06699186
Title: The Effects of Sleep After Delayed-onset Muscle Soreness, a Comparative Study
Brief Title: Sleep and Delayed-onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gülşah ÖZSOY, PhD, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SELCUKU_PT_GO_PAIN_001
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Delayed-onset Muscle Soreness; Sleep; Pain
Keywords: Acute Pain; Musculoskeletal Pain; Pain Threshold; Range of Motion; Sleep Deprivation
MeSH Terms: conditions — Pain; Acute Pain; Musculoskeletal Pain; Sleep Deprivation | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomised, single-blind, controlled trial. The patients were divided into two groups, designated as the "sleep group" and the "non-sleep group," through the implementation of a matched randomization method that considered both gender and age as variables.
Who Masked: Investigator
Masking Description: Prior to and following the interventions, all assessments were evaluated by a researcher who was blinded to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Group (Experimental): The sleep group was instructed to engage in a minimum of six hours of sleep over the course of the 24-hour observation period. Individuals who slept for a duration of less than six hours were excluded from the study.
  Interventions: Other: Sleep
- Non-sleep group (Active Comparator): The participants were permitted to sleep for a maximum of four hours in total over the course of the 24-hour period in non-sleep group.
  Interventions: Other: Non-sleep

INTERVENTIONS:
Other: Sleep — A training programme was devised which involved the participants performing maximum squat repetitions with their own body weight as a workload, in order to induce delayed-onset muscle soreness in the quadriceps. Before the maximum squat repetition, all participants performed a warm-up programme including 5 minutes of walking. Participants were instructed to perform the maximum number of repetitions within the one minute allotted for each set of squats and, after a 10-second rest period, to continue the programme in the same cycle until exhaustion. In the initial 24-hour period following the intervention, participants were instructed to maintain their habitual sleep schedules. In consideration of the delayed-onset muscle soreness, which typically occurs between 24 to 48 hours following maximal squat intervention.The sleep group was instructed to engage in a minimum of six hours of sleep over the course of the 24-hour observation period.
  Arms: Sleep Group
Other: Non-sleep — A similar delayed-onset muscle soreness inducing protocol was applied to the sleep group.Participants in the non-sleep group were subjected to sleep restriction. The participants were permitted to sleep for a maximum of four hours in total over the course of the 24-hour period in non-sleep group.
  Arms: Non-sleep group

SUMMARY:
There is a need for further experimental research in order to gain a more in-depth understanding of this vicious cycle of pain and sleep disorders. Although the effects of chronic pain and its impact on sleep have been extensively researched, the influence of sleep on acute pain has been addressed in only a limited number of studies. A more comprehensive grasp of the manner in which sleep influences the pain sensory profile subsequent to an acute injury may offer insight into the significance of sleep during recovery stage. In this respect, the objective of this study was to examine the effect of sleep on pain perception, pain sensitivity and range of motion following the induction of delayed onset muscle soreness (DOMS) through eccentric loading, specifically through the performance of squat exercises.

DETAILED DESCRIPTION:
Delayed onset muscle soreness (DOMS) represents a phenomenon characterised by a range of symptoms, encompassing varying degrees of muscle stiffness and pain, from mild to severe, with the potential to cause considerable functional impairment. This may be attributed to muscle damage and subsequent inflammation resulting from eccentric contractions or activities of an unusually intense nature. In accordance with these principles, exercise-induced DOMS typically manifests following an abrupt increase in exercise intensity, the execution of unconventional exercise movements, and most notably, following the performance of exercises that necessitate eccentric muscle actions . DOMS frequently results in a reduction in muscle function, including a decline in strength, a narrowing of the range of motion, increased pain sensitivity, and a decrease in the intensity of proprioception sensations within a period of 24 to 72 hours, with the potential for these effects to persist for several days. The processes underlying of DOMS comprise overstretching of sarcomeres, mechanical stresses in muscle structures, overlaps and disruption of filaments, and reactions of biochemical that affect contractile structures of muscle. Furthermore, inflammatory processes linked to oxidative stress and an increased pain receptors sensitivity is additional factors contributing to the development of DOMS .

One of the most significant factors affecting pain is sleep. Those suffering from persistent pain consistently indicate inferior sleep quality in comparison to controls , and a direct correlation has been observed between the quality of sleep and the severity of pain experienced by individuals. It is established in the literature that the sensitisation of pain mechanisms is raised in both intervention models of acute pain and chronic pain. Furthermore, individuals who experience primary insomnia without pain report heightened sensitivity to pain and an increased frequency of spontaneous pain episodes compared to control subjects. The findings of experimental studies indicate that sleep disruption in healthy individuals is linked to a considerable rise in pain sensitivity, potentially associated with elevated serum concentrations of pro-inflammatory biomarkers, even in the absence of tissue damage. This results in a vicious cycle of pain and sleep disorders, with each condition precipitating the other, thereby rendering the problem challenging to comprehend.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic individuals
* Aged 18-25 years

Exclusion Criteria:

* Those who have functional exercise restrictions,
* Those with chronic cardiac or pulmonary diseases such as chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease and heart failure that may affect respiratory muscle strength and respiratory functions,
* Those with orthopedic problems, persistent neck and back pain and/or radiculopathy that prevent them from participating in the study,
* Those with diagnosed psychiatric disorders,
* Participants with cooperation problems that may prevent evaluations and treatment will not be included in the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
The pressure pain thresholds | 2 days
  The pressure pain thresholds (PPT) were recorded at two pre-defined locations (tibialis anterior and quadriceps) using an electronic digital display algometer (Commander Echo® Algometer, JTECH Medical) with a 1-cm² probe. The tibialis region was measured by positioning the tibialis anterior muscle at a distance of 8 cm from the tibial tuberosity along a line extending from the tibial tuberosity to the lateral malleolus. For the quadriceps region, the measurement was made on the rectus femoris muscle at the point between the base of the patella and the anterior superior iliac spine.
Numeric pain rating scale | 2 days
  The presence of DOMS was evaluated using a numeric pain rating scale (NPRS) with a range of 0 to 10. The participants were informed of the scale, which ranged from 0 (no pain) to 10 (extreme pain), and were subsequently asked to report the corresponding pain sensation.
Range of motion evaluation | 2 days
  Range of motion evaluations were conducted through the assessment of knee and hip flexion using a universal goniometer
Pittsburgh Sleep Quality Index | 2 days
  The sleep status of the participants was evaluated using the Pittsburgh Sleep Quality Index (PSQI) and routine sleep duration

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ducas J, Memari S, Houle M, Schwendenmann Y, Abboud J, Yiou E, Descarreaux M. Impact of lumbar delayed-onset muscle soreness on postural stability in standing postures. Gait Posture. 2024 Mar;109:201-207. doi: 10.1016/j.gaitpost.2024.02.001. Epub 2024 Feb 8. PMID 38350184
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] da Silva W, Machado AS, Lemos AL, de Andrade CF, Priego-Quesada JI, Carpes FP. Relationship between exercise-induced muscle soreness, pain thresholds, and skin temperature in men and women. J Therm Biol. 2021 Aug;100:103051. doi: 10.1016/j.jtherbio.2021.103051. Epub 2021 Jul 11. PMID 34503798
- [Background] Farias-Junior LF, Browne RAV, Freire YA, Oliveira-Dantas FF, Lemos TMAM, Galvao-Coelho NL, Hardcastle SJ, Okano AH, Aoki MS, Costa EC. Psychological responses, muscle damage, inflammation, and delayed onset muscle soreness to high-intensity interval and moderate-intensity continuous exercise in overweight men. Physiol Behav. 2019 Feb 1;199:200-209. doi: 10.1016/j.physbeh.2018.11.028. Epub 2018 Nov 22. PMID 30471384
- [Background] Njeim P, Faust A, Casgrain J, Karelis AD, Boutros GH. Delayed Onset Muscle Soreness Following Acute Resistance Exercise in Untrained Females: A Comparative Study Between Vegans and Omnivores. Int J Sports Med. 2024 Dec;45(14):1099-1106. doi: 10.1055/a-2350-8681. Epub 2024 Jul 31. PMID 39084325